CLINICAL TRIAL: NCT06115486
Title: EXERT-BCH: Prospective Study of EXErcise Regimens After Treatment for Breast Cancer to Improve Hypertrophy
Brief Title: EXERT-BCH Exercise Regimen to Improve Muscle Mass After Treatment of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EXERT-BCH
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Breast Carcinoma in Situ; Breast Cancer Female
Keywords: Cancer; Carcinoma in Situ; Hypertrophy; Exercise
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Neoplasms; Carcinoma in Situ; Hypertrophy; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will include rolling block randomization of two groups of 15 participants in each group. The 6-12-25 arm will be enrolled first, followed by the ACSM arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm / ACSM Guidelines (Other): The control group will follow resistance training guidelines from the American College of Sports Medicine (ACSM) with the goal of promoting hypertrophy
  Interventions: Other: Control Arm ACSM Guidelines
- Experimental Arm / EOC Guidelines (Experimental): The experimental group will use a regimen that is often used by strength and conditioning coaches to maximize hypertrophy, and is part of the standard regimens at the Exercise Oncology Center (EOC)
  Interventions: Other: Experimental Arm 6-12-25 repetitions per set

INTERVENTIONS:
Other: Control Arm ACSM Guidelines — The control group will follow resistance training guidelines from the American College of Sports Medicine. Eight to ten multi-joint exercises will be performed to stress the major muscle groups.
  Arms: Control Arm / ACSM Guidelines
Other: Experimental Arm 6-12-25 repetitions per set — The exercise regimens will employ a mixture of compound exercises utilizing both open and closed kinetic chain movements (CKC), focusing on exercises with the goal of increasing skeletal muscle mass and body composition. The regimen will incorporate 6, then 12, then 25 repetitions in sequence per set per muscle group with minimal amounts of rest between.
  Arms: Experimental Arm / EOC Guidelines

SUMMARY:
The purpose of this research study is to evaluate the outcomes of two standard of care group exercise regimens to increase muscle mass in women who have been treated with breast cancer.

DETAILED DESCRIPTION:
This protocol seeks to analyze patient outcomes of two standard of care, time-efficient, monitored group exercise regimens of high-load resistance training to improve hypertrophy in women who have been treated for ductal carcinoma in situ or invasive carcinoma of the breast.

As part of the standard exercise program, patients will undergo a fitness evaluation at the AHNCI Exercise Oncology and Resiliency Center before the start of the exercise program. This evaluation will be used to customize the patient exercise program. The exercise program consists of small group training sessions held approximately 3 times per week at the center for 12 weeks (3 months). The fitness evaluation and exercise program are standard of care. Participation in this study will last the duration of the exercise program, about 3 months. All group exercise sessions will be closely monitored by the center staff who are Certified Strength and Conditioning Specialists (CSCS).

ELIGIBILITY:
Inclusion Criteria:

Age 20-89 years

* Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast
* Women must have undergone treatment for breast cancer, including one or more of the following: surgery, radiation therapy, chemotherapy, immunotherapy, or hormonal therapy. Women undergoing active chemotherapy are not allowed on study. Immunotherapy or targeted agent usage is allowed.

Exclusion Criteria:

* Any current treatment with cytotoxic chemotherapy for breast cancer
* Inability to safely engage in group sessions of resistance training as deemed by study PI
* Severe arthritic, joint, cardiovascular, or musculoskeletal condition deemed by PI to be unsafe to engage in resistance training

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of all races/ethnicities
Enrollment: 30 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Determine changes in muscle and fat mass during and after each exercise regimen | The exercise program will last for 8 weeks and continuously monitored by the PI and clinical team.
  The experimental group will follow a 6-12-25 program geared at optimizing hypertrophy and metabolism via high volume and increased time under tension.

SECONDARY OUTCOMES:
Determine adherence defined as number of sessions attended of total sessions | The exercise program will last for 8 weeks and continuously monitored by the PI and clinical team.
  The experimental group will follow a 6-12-25 program geared at optimizing hypertrophy and metabolism via high volume and increased time under tension.
Determine changes in strength measured via load calculations (repetitions x sets x weight) | The exercise program will last for 8 weeks and continuously monitored by the PI and clinical team.
  The experimental group will follow a 6-12-25 program geared at optimizing hypertrophy and metabolism via high volume and increased time under tension.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD, CSCS, Principal Investigator — Radiation Oncologist
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data